CLINICAL TRIAL: NCT04278703
Title: The Utilization of Opioid Medication Following ACL Reconstruction
Brief Title: Opioids Following ACL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020 TJ 03
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Oxycodone

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 15 opioid tablets perscribed (Active Comparator): For this treatment arm, patients will be given a prescription of 15 tablets of Oxycodone which they may take to alleviate post-operative pain
  Interventions: Drug: Oxycodone
- 25 opioid tablets perscribed (Active Comparator): For this treatment arm, patients will be given a prescription of 15 tablets of Oxycodone which they may take to alleviate post-operative pain
  Interventions: Drug: Oxycodone
- 35 opioid tablets perscribed (Active Comparator): For this treatment arm, patients will be given a prescription of 15 tablets of Oxycodone which they may take to alleviate post-operative pain
  Interventions: Drug: oxycodone

INTERVENTIONS:
Drug: Oxycodone — Patients will be given a prescription for 15 opioid tablets for post-operative pain
  Arms: 15 opioid tablets perscribed
Drug: Oxycodone — Patients will be given a prescription for 25 opioid tablets for post-operative pain
  Arms: 25 opioid tablets perscribed
Drug: oxycodone — Patients will be given a prescription for 35 opioid tablets for post-operative pain
  Arms: 35 opioid tablets perscribed

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a post-operative opioid pain 18 management protocol for anterior cruciate ligament reconstruction (ACLR).

ELIGIBILITY:
Inclusion Criteria:

- All patients undergoing primary ACLR for ACL tear, including patients with concomitant 76 meniscectomy or meniscal repair.

Exclusion Criteria:

* Concomitant procedure other than meniscectomy or meniscal repair.
* ACL revision
* History of chronic pre-operative opioid use
* History of substance abuse
* Workmen's compensation claims
* Pregnancy

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2019-02-15 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain | 14 days post-operative
  Post-operative pain as reported by patients on a 0-10 VAS pain scale. 0 is no pain and 10 is worst pain imaginable

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedics at Egg Harbor Township, Egg Harbor, New Jersey, United States